CLINICAL TRIAL: NCT06413251
Title: Boxing Training Effects on Cardiovascular Risk, Quality of Life, Endothelial Function, and Blood Flow Patterns in Individuals With Elevated Blood Pressure or Stage 1 Hypertension
Brief Title: Clinical Effectiveness of Boxing Training in Individuals With Elevated Blood Pressure or Stage 1 Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1364179-3
Record Dates: First submitted 2023-11-22; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Elevated Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from the University of Texas at El Paso and its surroundings. They will be identified by a preliminary blood pressure screening and a health questionnaire. The inclusion criteria will consist on: (1) ≥18 years old, (2) SBP between 120-139 mmHg or DBP between 80-89 mmHg obtained from 2 different days, (3) an estimated 10-year risk of CVD ≤10%, calculated by the ACC/AHA Pooled Cohort Equations, and (4) no current participation in 3 or more days per week of endurance or resistance exercise training. Exclusion criteria will include non-controlled cardiac, pulmonary, or metabolic diseases, smoking, consumption of nutritional supplements containing antioxidants, and any physical impairment to exercise.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boxing (Experimental): The boxing training intervention will consist of three exercise sessions per week on nonconsecutive days for six weeks
  Interventions: Other: Boxing Training
- Control (Placebo Comparator): The control group will perform three days per week 10 minutes a flexibility intervention.
  Interventions: Other: Control flexibility

INTERVENTIONS:
Other: Boxing Training — The boxing training intervention will consist of three exercise sessions per week on nonconsecutive days for six weeks. Participants will be instructed to complete 10 rounds of three minutes with a one-minute resting period interspersed. Four rounds will consist of heavy bag punching (e.g. straight, jab, hook) at 60% VO2max and three rounds at 90-95% VO2max, while the remaining 3 rounds will be focused on mitt work at 60% VO2max.
  Other Names: Exercise
  Arms: Boxing
Other: Control flexibility — The control group will perform three days per week 10 minutes of dynamic articular movement, five minutes of uni pedal stance, and five minutes of stretching of the upper limbs for six weeks.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to determine whether boxing training reduces cardiovascular risk in elevated blood pressure or hypertension stage 1 individuals.

The main questions it aims to answer are (1) if boxing training reduces peripheral and central blood pressure and (2) if boxing training improves cardiovascular function in elevated blood pressure or hypertension stage 1 individuals.

Participants with elevated blood pressure or hypertension stage 1 will be randomly divided into a control group or an intervention group. The latter group will be involved in boxing training, 3 days per week for 6 weeks.

Researchers will compare clinical and cardiovascular outcomes between the control and the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* Systolic blood pressure between 120-139 mmHg and/or diastolic blood pressure between 80-89 mmHg obtained from 2 different days.
* an estimated 10-year risk of CVD ≤10%, calculated by the ACC/AHA Pooled Cohort Equations.
* no current participation in 3 or more days per week of endurance or resistance exercise training.

Exclusion Criteria:

* non-controlled cardiac, pulmonary, or metabolic diseases.
* smoking, consumption of nutritional supplements containing antioxidants.
* any physical impairment to exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline brachial blood pressure after week six | pre-intervention and immediately after the intervention
  Resting systolic and diastolic blood pressure (mmHg)

SECONDARY OUTCOMES:
Central Blood Pressure | pre-intervention and immediately after the intervention
  Pulse wave analysis (mmHg)
Vascular function | pre-intervention and immediately after the intervention
  Flow mediated dilation (%)
Plethysmography | pre-intervention and immediately after the intervention
  Forearm and Calf Blood Flow (ml/min/100 ml tissue)
Maximum Oxygen Uptake | pre-intervention and immediately after the intervention
  Cardiopulmonary Test (ml/kg/min)
Nitric Oxide Bioavailability | pre-intervention and immediately after the intervention
  Blood Biomarker NOx (μmol/L)
Body Fat Percentage | pre-intervention and immediately after the intervention
  Dual energy x-ray absorptiometry Scan to assess Body Fat %
Lean Mass | pre-intervention and immediately after the intervention
  Dual energy x-ray absorptiometry Scan to assess lean mass (kg)
Quality of Life measured by the short-form 36 (SF-36) | pre-intervention and immediately after the intervention
  The short form 36 (SF-36) is a short survey that covers a total of 8 sub-dimensions related to physical and mental health: (1) Physical Functioning, (2) Role Limitations due to Physical Problems, (3) Social Functioning, (4) Bodily Pain, (5) General Mental Health, (6) Role Limitations due to Mental Problems, (7) Vitality, and (8) General Health Perceptions. The SF-36 includes a diverse mixture of continuous item scaling methods and is comprised of 10 items with balanced multi-item response formats (range from 1 to 5), 7 items with a dichotomous response format (1 or 2), and 19 items with non-balanced multi-item response formats (nine items range from 1 to 3 and ten items range from 1 to 6). To obtain the raw score for each sub-dimension, 10 items are reversed. Then, raw values for each sub-dimension are summed. Finally, the raw scores are transformed to a 0-to-100 scale for each sub-dimension. Higher scores indicate higher Quality of Life from 0 (worst) to 100 (best).
Arterial Stiffness | pre-intervention and immediately after the intervention
  Pulse wave velocity from carotid to femoral artery (m/s)
C Reactive Protein (CRP) to assess inflammation | pre-intervention and immediately after the intervention
  Blood Biomarker CRP (mg/L)
Interleukin-6 (IL-6) to assess inflammation | pre-intervention and immediately after the intervention
  Blood Biomarker IL-6 (pg/ml)
Tumor necrosis factor alfa (TNFα) to assess inflammation | pre-intervention and immediately after the intervention
  Blood Biomarker TNFα (pg/ml)
8-isoprostane to assess inflammation | pre-intervention and immediately after the intervention
  Blood Biomarker 8-isoprostane (pg/ml)
Superoxide dismutase (SOD) to assess oxidative stress | pre-intervention and immediately after the intervention
  Blood Biomarker SOD (mU/ml)
Total Antioxidant Capacity (TAC) to assess oxidative stress | pre-intervention and immediately after the intervention
  Blood Biomarker TAC (mM/ml)
Lipid Profile | pre-intervention and immediately after the intervention
  Blood Biomarkers HDL-C, LDL-C, and total cholesterol (mg/dl)
Weight | pre-intervention and immediately after the intervention
  Weight in kilograms
Height | pre-intervention and immediately after the intervention
  Height in meters

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Only the PI will analyze the collected data.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT06413251/Prot_SAP_ICF_000.pdf